CLINICAL TRIAL: NCT05605535
Title: A Phase 2, Double-Blind, Placebo-Controlled, Multicenter Clinical Trial Comparing Chemoimmunotherapy (Paclitaxel-Carboplatin-Oregovomab) Versus Chemotherapy (Paclitaxel-Carboplatin-Placebo) as Neoadjuvant Therapy in Patients With Advanced Epithelial Ovarian, Fallopian Tube or Peritoneal Carcinoma
Brief Title: Oregovomab Plus Chemotherapy in Neo-adjuvant Setting in Newly Diagnosed Patients With Advanced Epithelial Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CanariaBio Inc. (Industry)
Collaborators: Raptim Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QPT-ORE-006
Record Dates: First submitted 2022-10-25; First posted 2022-11-04 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Neoplasm Epithelial; Ovarian Cancer; Fallopian Tube Neoplasms; Peritoneal Carcinoma; Ovarian Serous Adenocarcinoma
Keywords: Ovarian cancer; Phase 2; Oregovomab; Chemoimmunotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — oregovomab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination of Oregovomab and chemotherapy (Experimental): Six (6) cycles of chemotherapy with oregovomab given only at specific cycles (Cycle 1, Cycle 3, Cycle 4, Cycle 6 and Cycle 6 plus 12 weeks).
  Interventions: Biological: Oregovomab; Drug: Paclitaxel; Drug: Carboplatin
- Combination of Placebo and chemotherapy (Placebo Comparator): Six (6) cycles of chemotherapy with placebo given only at specific cycles (Cycle 1, Cycle 3, Cycle 4, Cycle 6 and Cycle 6 plus 12 weeks).
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Biological: Placebo

INTERVENTIONS:
Biological: Oregovomab — 2 mg, dissolved in 2 mL of 0.9% Sodium Chloride Injection USP, then added to 50 mL of Sodium Chloride Injection USP infused over 20 ± 5 minutes
  Other Names: MAb-B43.13
  Arms: Combination of Oregovomab and chemotherapy
Drug: Paclitaxel — 175 mg/m^2, every 3 weeks
  Other Names: Taxol
Drug: Carboplatin — AUC 5 or 6 IV Day 1 x 6 cycles (every 21 days)
  Other Names: Paraplatin
Biological: Placebo — 2 mg, dissolved in 2 mL of 0.9% Sodium Chloride Injection USP, then added to 50 mL of Sodium Chloride Injection USP infused over 20 ± 5 minutes
  Arms: Combination of Placebo and chemotherapy

SUMMARY:
A clinical study to compare the efficacy and safety of five administrations of oregovomab versus placebo, infused in schedule dependent sequence with specific cycles of a standard six-cycle chemotherapy regimen (paclitaxel and carboplatin), for the treatment of patients with newly diagnosed advanced ovarian cancer who are planned to receive neoadjuvant treatment followed by interval debulking surgery (IDS) and adjuvant treatment.

DETAILED DESCRIPTION:
Phase 2, double-blind, placebo-controlled, multi-center study to compare the efficacy and safety of five administrations of oregovomab 2 mg IV versus placebo, infused in a schedule dependent sequence with specific cycles of a standard six-cycle chemotherapy regimen (paclitaxel and carboplatin), for the treatment of patients with newly diagnosed advanced ovarian cancer who are planned to receive neoadjuvant treatment. Patients will receive oregovomab or placebo at Cycles 1 and 3 in combination with paclitaxel and carboplatin prior to IDS, followed by oregovomab or placebo at Cycles 4 and 6 in combination with paclitaxel and carboplatin, and oregovomab or placebo monotherapy at Cycle 6 plus 12 weeks.

This study will screen approximately 96 patients to randomize approximately 88 patients. All eligible patients will be stratified by FIGO Stage (Stages IIIA, IIIB versus Stages IIIC, IV).

The study includes screening period, treatment period, post-treatment follow up, safety follow and long term follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Adult females 18 years old or older.
2. Newly diagnosed epithelial adenocarcinoma of ovarian, fallopian tube or peritoneal origin FIGO Stage III or IV patients whose disease is confirmed based on biopsy sample.
3. Eligible histologic epithelial cell types: high grade serous adenocarcinoma, high grade endometrioid adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, or adenocarcinoma not otherwise specified (N.O.S.).
4. Suitable venous access for the study-required procedures.
5. Serum CA125 levels ≥ 50 U/mL prior to Cycle 1 of NACT chemotherapy + oregovomab or placebo.
6. Adequate bone marrow function:

   1. Absolute neutrophil count (ANC) ≥ 1,500/μL.
   2. Platelets ≥100,000/μL.
   3. Hemoglobin ≥ 8.0 g/dL (Note: Blood transfusion is permitted up to 48 hours before the first dose of study treatment).
7. Adequate liver function:

   1. Bilirubin < 1.5 times upper limit normal (ULN).
   2. SGOT/AST and SGPT/ALT < 2.5 times ULN.
8. Adequate renal function:

   a. Creatinine ≤ 1.5 times ULN.
9. ECOG Performance Status of 0, 1 or 2.
10. Women of childbearing potential must be willing to avoid pregnancy by using a highly effective method of contraception from the first dose of study treatment to 6 months after last dose of study treatment.
11. Signed written informed consent form and authorization permitting release of personal health information. Ability to comply with treatment and follow up

Exclusion Criteria:

1. Patients with mucinous adenocarcinoma, carcinosarcoma, tumors with neuroendocrine features and low-grade adenocarcinoma (including low grade serous and FIGO grade 1 endometrioid adenocarcinomas of the ovary).
2. FIGO Stage IV patients:

   1. FIGO stage IV patients suspected or diagnosed with bone or brain metastasis are excluded.
   2. FIGO stage IV patients diagnosed with lung and/or liver metastasis with tumour size more than 2 cm are excluded.
   3. FIGO stage IV patients diagnosed with lung and/or liver metastasis and expected to administer with more than 3 cycles of chemotherapy and/or not suitable for interval debulking surgery are excluded.
3. Patients must not have received any prior chemotherapy, immunotherapy, targeted or hormonal therapy.
4. Patients who are lactating and breastfeeding or have a positive serum pregnancy test within 14 days prior to the first dose of study treatment.
5. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study treatment according to this protocol.
6. Active autoimmune disease such as rheumatoid arthritis, SLE, ulcerative colitis, Crohn's Disease, MS, or ankylosing spondylitis, requiring active disease modifying treatment.
7. Known allergy to murine proteins or hypersensitivity to any of the excipients of the oregovomab, paclitaxel, or carboplatin.
8. Chronically treated with immunosuppressive drugs such as cyclosporine, adrenocorticotropic hormone (ACTH), etc.
9. Chronic therapeutic corticosteroid use, defined as > 5 days of prednisone or equivalent, except for inhalers or those on a pre-planned steroid taper. (Note: Premedication with corticosteroids per institutional standard of care is allowed.)
10. Recognized acquired, hereditary, or congenital immunodeficiency disease, including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia.
11. Clinically significant active infection(s) at the time of screening.
12. Any of the following conditions (on-study testing is not required):

    1. Known HIV-infected patients unless on effective anti-retroviral therapy with an undetectable viral load within 6 months prior to randomization, or
    2. Known or suspected hepatitis B if active infection (patients with chronic hepatitis B infection must have an undetectable HBV viral load on suppressive therapy, if indicated; positive surface antibody alone is not an exclusion), or
    3. Known or suspected hepatitis C infection which has not been treated and cured unless currently on treatment with an undetectable viral load.
13. Uncontrolled or life-threatening diseases compromising safety evaluation. Diagnosed or treated for another malignancy within 5 years before the first dose, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer, ductal carcinoma in-situ (DCIS) of the breast or cervix carcinoma in situ are not excluded if they have undergone complete resection. a. Synchronous endometrial cancer, but a prior diagnosis of endometrial cancer within 5 years is not excluded if all of the following conditions are met: Stage IA, superficial myometrial invasion, without lymphovascular invasion, and not poorly differentiated subtypes including papillary serous, clear cell or other FIGO Grade II and III lesions.

15. Contraindication to the use of pressor agents. 16. Undergone prior surgical debulking. 17. History or evidence upon physical examination of CNS disease, seizures not controlled with standard medical therapy, or any brain metastases. 18. Any of the following cardiovascular conditions:

1. Acute myocardial infarction within 6 months before the first dose of study treatment.
2. Current history of New York Heart Association (NYHA) Class III or IV heart failure
3. Evidence of current uncontrolled cardiovascular conditions including cardiac arrhythmias, angina, pulmonary hypertension, or electrocardiographic clinically significant findings. 19. Unable to read or understand or unable to sign the necessary written consent before starting treatment. 20. May not receive any live, attenuated vaccine administered within 28 days (or 4 weeks) prior to enrollment, during the study, and for at least 90 days after the last dose of study treatment. 21. Patients who will receive Hyperthermic Intraperitoneal Chemotherapy (HIPEC), any other anti-cancer medications, including bevacizumab, PARPi, or any other investigational agent(s) with 3 cycles of paclitaxel and carboplatin neo-adjuvant treatment will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women 18 years of age and older
Enrollment: 88 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) Rate at 12 months | At 12 months
  PFS, is assessed from date of randomization to the date of first documented progression as per RECIST v1.1 as determined by the investigator or death due to any cause.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | At 3 months
  Overall response rate is defined according to RECIST v1.1 measured at end of first 3 cycles of study treatment and prior to debulking surgery treatment:
  * Complete response
  * Partial Response
Disease Control Rate (DCR): | At 3 months
  Disease control rate is defined according to RECIST v1.1 measured at end of first 3 cycles of treatment and prior to debulking surgery treatment:
  * Complete response
  * Partial Response
  * Stable Disease
Response to Surgery | At 4 months
  Upon completion of neo-adjuvant treatment and IDS, Response to surgery will be assessed on the size of residual disease - none (R0), < 1 cm (R1), ≥ 1 cm (R2)
Progression Free Survival | Approximately up to 4 years
  Progression free survival is defined as date of randomization to date of first documented progression as per RECIST v1.1 as determined by the investigator or death due to any cause and OS defined as date of randomization to date of death due to any cause.
Overall Survival | Approximately up to 8 years
  Overall survival is defined as date of randomization to date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jada Srinivasa Rao, PhD, Study Director — CanariaBio Inc.
Locations (14):
- India (14):
  - Omega Hospitals, Visakhapatnam, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Himalaya Cancer Hospital and Research Institute, Vadodara, Gujarat
  - Kailash Cancer Hospital and Research Centre, Vadodara, Gujarat
  - KLES Dr. Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Regional Cancer Centre, Medical College, Trivandrum, Kerala
  - Sri Ram Cancer Hospital, Jaipur, Rajasthan
  - Saveetha Medical College and Hospitals, Chennai, Tamil Nadu
  - Sri Ramchandra Medical Centre, Chennai, Tamil Nadu
  - MNJ Cancer Hospital, Hyderabad, Telangana
  - King Georges Medical University, Lucknow, Uttar Pradesh
  - Institute of Medical Sciences, BHU, Varanasi, Uttar Pradesh
  - JIPMER, Puducherry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brewer M, Angioli R, Scambia G, Lorusso D, Terranova C, Panici PB, Raspagliesi F, Scollo P, Plotti F, Ferrandina G, Salutari V, Ricci C, Braly P, Holloway R, Method M, Madiyalakan M, Bayever E, Nicodemus C. Front-line chemo-immunotherapy with carboplatin-paclitaxel using oregovomab indirect immunization in advanced ovarian cancer: A randomized phase II study. Gynecol Oncol. 2020 Mar;156(3):523-529. doi: 10.1016/j.ygyno.2019.12.024. Epub 2020 Jan 6. PMID 31916979
- [Background] Braly P, Nicodemus CF, Chu C, Collins Y, Edwards R, Gordon A, McGuire W, Schoonmaker C, Whiteside T, Smith LM, Method M. The Immune adjuvant properties of front-line carboplatin-paclitaxel: a randomized phase 2 study of alternative schedules of intravenous oregovomab chemoimmunotherapy in advanced ovarian cancer. J Immunother. 2009 Jan;32(1):54-65. doi: 10.1097/CJI.0b013e31818b3dad. PMID 19307994
- [Background] Berek J, Taylor P, McGuire W, Smith LM, Schultes B, Nicodemus CF. Oregovomab maintenance monoimmunotherapy does not improve outcomes in advanced ovarian cancer. J Clin Oncol. 2009 Jan 20;27(3):418-25. doi: 10.1200/JCO.2008.17.8400. Epub 2008 Dec 15. PMID 19075271